CLINICAL TRIAL: NCT06156995
Title: Clinical Study on the Treatment of Colonic Slow Transit Constipation by Deep Acupuncture at Zhongliao Point Stimulating Sacral Nerve
Brief Title: Deep Needling at Zhongliao Point to Stimulate the Sacral Nerve for the Treatment of Slow Transit Constipation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guoliang Wu (Other)
Collaborators: Qianfoshan Hospital (Other)
Responsible Party: Sponsor-Investigator, Guoliang Wu, Principal Investigator, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GlWu
Record Dates: First submitted 2023-11-18; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Constipation
Keywords: Constipation
MeSH Terms: conditions — Constipation | interventions — mosapride

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Using 0.30mm × 75mm millineedle (produced by Suzhou Medical Equipment Factory, Huatuo brand) deeply punctures the Zhongliao acupoint to reach the sacral nerve. The acupuncture needle is connected using the MuhiStim Sensor nerve stimulator produced by Pajunk in Germany. Connect the positive pole to the left Zhongliao hole and the negative pole to the right Zhongliao hole. The frequency, current, and pulse width of sacral nerve electrical stimulation are 2 Hz, 5mA, and 0.1 ms, respectively.Electroacupuncture stimulates the sacral nerve for 30 minutes, once a day, five times a week. After the treatment, rest for two days before starting the next treatment. Five sessions are considered as one course of treatment, with a total of four courses for four consecutive weeks.
  Interventions: Device: Deep Acupuncture at Zhongliao Point to Stimulate Sacral Nerve
- control group (Active Comparator): Mosapride citrate tablets (produced by Lunan Beite Pharmaceutical Co., Ltd., with the national drug approval number H19990317), oral administration, 5mg once, three times a day, taken before meals. 5 days is one course of treatment, with 2 days of rest during the treatment period. The total treatment period is 4 weeks, with a total of 4 courses.
  Interventions: Drug: Oral Mosapride Tablets

INTERVENTIONS:
Device: Deep Acupuncture at Zhongliao Point to Stimulate Sacral Nerve — Using 0.30mm × 75mm millineedle (produced by Suzhou Medical Equipment Factory, Huatuo brand) deeply punctures the Zhongliao acupoint to reach the sacral nerve. The acupuncture needle is connected using the MuhiStim Sensor nerve stimulator produced by Pajunk in Germany. Connect the positive pole to the left Zhongliao hole and the negative pole to the right Zhongliao hole. The frequency, current, and pulse width of sacral nerve electrical stimulation are 2 Hz, 5mA, and 0.1 ms, respectively.Electroacupuncture stimulates the sacral nerve for 30 minutes, once a day, five times a week. After the treatment, rest for two days before starting the next treatment. Five sessions are considered as one course of treatment, with a total of four courses for four consecutive weeks.
  Arms: Treatment group
Drug: Oral Mosapride Tablets — Mosapride citrate tablets (produced by Lunan Beite Pharmaceutical Co., Ltd., with the national drug approval number H19990317), oral administration, 5mg once, three times a day, taken before meals. 5 days is one course of treatment, with 2 days of rest during the treatment period. The total treatment period is 4 weeks, with a total of 4 courses.
  Arms: control group

SUMMARY:
Clinical Study on the Treatment of Colonic Slow Transit Constipation by Deep Acupuncture at Zhongliao Point Stimulating Sacral Nerve

DETAILED DESCRIPTION:
1. Observing the clinical efficacy of deep acupuncture at Zhongliao point to stimulate the sacral nerve in the treatment of slow transit constipation of the colon through changes in main research indicators such as defecation frequency, stool shape, and fecal weakness.
2. Clarify the technical focus and difficulties of deep needling at Zhongliao point to stimulate the sacral nerve in the treatment of colonic slow transit constipation, providing a basis for guiding clinical promotion and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meets the diagnostic criteria for Slow transit constipation deficiency of both qi and yin;
* Age 18-65 years old;
* I have not been treated with intestinal motility drugs in the past month.
* Those who have informed consent and voluntarily participate in signing an informed consent form, adhere to medical advice for treatment, and undergo regular follow-up visits.

Exclusion Criteria:

* Other Traditional Chinese Medicine Syndrome Differentiation Types of Constipation.
* Concomitant severe heart, lung, and kidney diseases, neurological diseases, and metabolic diseases;
* Discovering organic lesions such as colorectal cancer and colorectal hyperplasia through colonoscopy, abdominal pelvic CT, or barium enema;
* Patients with severe mental illness or mental illness or cognitive impairment.
* Children, pregnant women, lactating women, and pregnant women.
* Those who stop taking medication at will or use other medications on their own during treatment, do not follow medical advice for treatment, or have incomplete information that affects the judgment of results, safety, and efficacy.
* Have a history of abdominal surgery.
* History of needle sickness.
* People with a tendency to bleed.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Cleveland Constipation Score（CCS） | Each group of patients was evaluated for indicators 1 week before treatment, 4 weeks after treatment, and 8 weeks after treatment.
  The Clinical Scoring Scale for Constipation Patients (CCS) is mainly a scoring standard for quantifying the severity of constipation. Its content mainly includes 8 items: frequency of defecation, difficulty in defecation, feeling of incomplete defecation, abdominal pain, defecation time, type of help needed, frequency of difficulty in resolving constipation every 24 hours, and duration of constipation. The score range is 0-30 points, and the higher the score, the more severe the constipation is.
Changes in the score of Bristol fecal trait scale | Each group of patients was evaluated for indicators 1 week before treatment, 4 weeks after treatment, and 8 weeks after treatment.
  Type 1 is a separated hard mass, type 2 is a clump shape, type 3 is a dry and cracked sausage shape, type 4 is a soft sausage shape, type 5 is a soft mass, type 6 is a mud shape, and type 7 is a watery stool. Each patient is assigned a score of 1-7. The patient confirms their stool classification based on the Bristol fecal trait scale and records it.

SECONDARY OUTCOMES:
Changes in the frequency of complete spontaneous bowel movements (CSBM) | Each group of patients was evaluated for indicators 1 week before treatment, 4 weeks after treatment, and 8 weeks after treatment.
  Complete spontaneous bowel movement (CSBM) refers to the number of times a patient can spontaneously defecate and feel completely discharged every week without taking remedial laxatives or manual assistance;Observation indicators are mainly based on the defecation record card provided by the patient.
Changes in the frequency of spontaneous bowel movements (SBM) | Each group of patients was evaluated for indicators 1 week before treatment, 4 weeks after treatment, and 8 weeks after treatment.
  Spontaneous bowel movement (SBM) refers to the number of times a patient spontaneously defecates per week, including feeling exhausted and feeling unable to defecate. Observation indicators are mainly based on the defecation record card provided by the patient.
Changes in the Quality of Life Scale (PAC-QOL) scores of patients with constipation | Each group of patients was evaluated for indicators 1 week before treatment, 4 weeks after treatment, and 8 weeks after treatment.
  The international constipation patient quality of life rating scale designed based on PROs is mainly a survey questionnaire for the quality of life of constipation patients. Patients are scored before and after treatment, and physicians collect and record their individual and total scores for physical discomfort, psychological discomfort, constipation related anxiety, and satisfaction with treatment. The score is 0-112 points, and the higher the score, the worse the quality of life.
Incidence of the adverse reactions | Each group of patients was evaluated for indicators 1 week before treatment, 4 weeks after treatment, and 8 weeks after treatment.
  The acupuncture operator records the adverse reactions of the patient after the acupuncture operation (such as dizziness, infection, pelvic organ and nerve damage, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Pang jing, M.D., Principal Investigator — Qianfoshan Hospital
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No